CLINICAL TRIAL: NCT06831981
Title: Radiochemotherapy With Concomitant Deep Regional Hyperthermia in Locally Advanced Rectal Cancer. A Prospective, Randomized Phase III Trial.
Brief Title: Hyperthermia With Chemoradiotherapy in Rectal Cancer
Acronym: ARO 2024-13
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University Hospital Erlangen (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 182/2024BO1
Record Dates: First submitted 2024-12-03; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-11

CONDITIONS: Rectal Cancer
Keywords: Hyperthermia; TME; high risk rectal tumors; locally advanced retal cancer; total neoadjuvant therapy; organ preservation
MeSH Terms: conditions — Rectal Neoplasms; Hyperthermia | interventions — Diathermy; Radiotherapy; Drug Therapy; Fluorouracil; Consolidation Chemotherapy; Folfox protocol

STUDY DESIGN:
Intervention Model Description: Radiochemotherapy of rectal cancer with (group 1) or without hyperthermia (group 2). Followed by consolidation chemotherapy (six courses). Option for 5x5 short time radiotherapy without hyperthermia followed by nine courses of consolidation chemotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiochemotherapy with hyperthermia followed by consolidation chemotherapy (Experimental): Radiochemotherapy with hyperthermia followed by consolidation chemotherapy. After restaging decision to watch and wait in case of complete or near complete response or surgery
  Interventions: Other: Hyperthermia; Radiation: Radiotherapy; Drug: Chemotherapy with 5-fluorouracil; Drug: Consolidation chemotherapy with FOLFOX
- Radiochemotherapy without hyperthermia followed by consolidation chemotherapy (Active Comparator): Radiochemotherapy without hyperthermia followed by consolidation chemotherapy. After restaging decision to watch and wait in case of complete response or surgery
  Interventions: Radiation: Radiotherapy; Drug: Chemotherapy with 5-fluorouracil; Drug: Consolidation chemotherapy with FOLFOX

INTERVENTIONS:
Other: Hyperthermia — Additional hyperthermia to radiochemotherapy regime in Arm 1 and radiochemotherapy without additional hyperthermia in Arm 2.
  Arms: Radiochemotherapy with hyperthermia followed by consolidation chemotherapy
Radiation: Radiotherapy — Radiotherapy of the pelvis
Drug: Chemotherapy with 5-fluorouracil — Chemotherapy with 5-flurouracil is given in parallel to radiotherapy
Drug: Consolidation chemotherapy with FOLFOX — Consolidation chemotherapy with 5-fluorouracil and oxaliplatin

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of deep regional hyperthermia in the context of radiochemotherapy followed by consolidation chemotherapy in locally advanced rectal cancer.

Questions it aims to answer are:

* Can surgery be avoided if the tumor completely regresses?
* How high is the Local re-growth rate
* Is the treatment safe?
* Assessment of the Quality of life
* Rate of sphincter-sparing surgery
* Pathological staging, tumor downstaging
* Assessment of continence during the course of therapy

Participants will:

Undergo radiochemotherapy with or without addition of hyperthermia (50:50 randomisation) followed by standard consolidation chemotherapy. After treatment response evaluation surgery or non-operative management takes place.

DETAILED DESCRIPTION:
In this prospective, randomized phase III trial "Radiochemotherapy with concomitant deep regional hyperthermia in locally advanced rectal cancer" trial it is hypothesized that with the addition of hyperthermia complete response rates can be further increased resulting in a higher number of patients who can omit surgery in favor of organ preservation and a surveillance protocol. Patients receive radiochemotherapy with 5-FU or capecitabine followed by standard consolidation chemotherapy with 5-FU/folinic acid/oxaliplatin or CAPOX. Hyperthermia will take place based on a 1:1 randomisation. After evaluation of treatment response in week 22 patients will either undergo surgical resection in case of residual tumor or non-operative management when a clinical complete response is seen or repeat evaluation after another 3 months in case of a near clinical complete response. In selected cases endoscopic procedures can be considered as an alternative to radical surgery.The primary objective of the study is to evaluate the efficacy of deep regional hyperthermia in the context of radiochemotherapy followed by consolidation chemotherapy in locally advanced rectal cancer. As the primary endpoint TME-free survival will be used (TMEFS).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with histologically confirmed diagnosis of rectal cancer localized 0-12 cm from the anocutaneous line (i.e. lower and middle third of the rectum)
* Indication for total neoadjuvant therapy irrespective of participation in the current study.
* Any MRI staged rectal cancer with one of the following high-risk features:

  * cT4
  * cN2 (see Appendix)
  * Distance to mesorectal fascia 1mm or less.
  * Involved Lateral pelvic lymph nodes
  * EMVI (extramural venous invasion) positivity
* Staging requirements: High-resolution, thin-sliced (i.e. 3mm) magnetic resonance imaging (MRI) of the pelvis is the mandatory local staging procedure.
* Cross-sectional imaging of the abdomen and chest to exclude distant metastases.
* Aged at least 18 years. No upper age limit.
* WHO/ECOG Performance Status ≤ 1
* Adequate hematological, hepatic, renal and metabolic function parameters
* Informed consent of the patient

Exclusion Criteria:

* Lower border of the tumor localised more than 12 cm from the anocutaneous line as measured by rigid rectoscopy
* Tumors with microsatellite instability ("MSI-High Tumors") and the possibility for treatment with immune checkpoint inhibition.
* Contraindication for hyperthermia such as metal implants or pacemakers
* Distant metastases (to be excluded by CT scan of the thorax and abdomen)
* Preexisting fecal incontinence for solid stool
* Prior antineoplastic therapy for rectal cancer
* Prior radiotherapy of the pelvic region
* Major surgery within the last 4 weeks prior to inclusion
* Subject pregnant or breastfeeding, or planning to become pregnant within 6 months after the end of treatment
* Subject (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment (adequate: oral contraceptives, intrauterine device or barrier method in conjunction with spermicidal jelly)
* Other concomitant antineoplastic therapy
* Serious concurrent diseases, including neurologic or psychiatric disorders (incl. dementia and uncontrolled seizures), active, uncontrolled infections, active, disseminated coagulation disorder
* Clinically significant cardiovascular disease (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 6 months before enrolment
* Prior or concurrent malignancy ≤ 3 years prior to enrolment in study (Exception: non-melanoma skin cancer or cervical carcinoma FIGO stage 0-1), if the patient is continuously disease-free
* Known allergic reactions on study medication
* Known dihydropyrimidine dehydrogenase deficiency
* Psychological, familial, sociological or geographical conditions potentially hampering compliance with the study protocol and follow-up schedule (these conditions should be discussed with the patient before registration in the trial)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2036-06-01 (Estimated); Study Completion 2037-03-01 (Estimated)

PRIMARY OUTCOMES:
Two-year TME-free survival (TMEFS) | From September 2024 until September 2036
  The primary objective of the study is to evaluate the efficacy of deep regional hyperthermia in the context of radiochemotherapy followed by consolidation chemotherapy in locally advanced rectal cancer. As the primary endpoint two-year TME-free survival will be used (TMEFS).

CONTACTS AND LOCATIONS:
Overall Officials: Cihan Gani, MD, Prof. Dr., Principal Investigator — University Hospital Tuebingen
Locations (2):
- Germany (2):
  - University Hospital, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg

IPD SHARING:
Plan to Share IPD: Undecided